CLINICAL TRIAL: NCT04985019
Title: A Validation Study of Mobile Virtual Reality-Based Self-Care and Exposure Therapy Contents for the Treatment of Panic Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Jooyoung Oh, Clinical Assistant Professor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3-2018-0292
Record Dates: First submitted 2021-07-26; First posted 2021-08-02 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Panic Disorder
MeSH Terms: conditions — Panic Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I (Prepectoral) (Experimental): VR treatment group Participants received the Self-Guided Virtual Reality-based Cognitive Behavioral Therapy for panic disorder.
  Interventions: Procedure: Arm I (Prepectoral); Other: Arm II (Subpectoral)
- II (Subpectoral) (No Intervention): Waiting list Participants in a waiting list.

INTERVENTIONS:
Procedure: Arm I (Prepectoral) — Participants followed the Self-Guided Virtual Reality-based Cognitive Behavioral Therapy for 4 weeks.
  Arms: I (Prepectoral)
Other: Arm II (Subpectoral) — Participants followed the Self-Guided Virtual Reality-based Cognitive Behavioral Therapy for 4 weeks.
  Arms: I (Prepectoral)

SUMMARY:
The purpose of this study is to determine whether mobile-based virtual reality exposure treatement can reduce the symptoms of panic disorder and the symptoms of depression and anxiety than the waitlist group

ELIGIBILITY:
Inclusion Criteria:

- Meet Diagnostic Statistical Manual criteria for panic disorder(with or without agoraphobia) .

No change in drug dosage during the study period

Exclusion Criteria:

- Patients with a history of major neurological or significant medical illness, or met the diagnostic criteria of current substance misuse

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2021-01-04 (Actual); Study Completion 2021-01-04 (Actual)

PRIMARY OUTCOMES:
The Panic Disorder Severity Scale | 4 weeks
  The Panic Disorder Severity Scale consists of 7 items, each rated on a 5-point scale that assesses panic frequency, distress during panic, panic-focused anticipatory anxiety, phobic avoidance of situations, phobic avoidance of physical sensations, impairment in work functioning, and impairment in social functioning

SECONDARY OUTCOMES:
The heart rate variability | 4 weeks
  The heart rate variability is the physiological recordings of the variation in the time interval between consecutive heartbeats in milliseconds
The Hamilton Rating Scale for Depression | 4 weeks
  The Hamilton Rating Scale for Depression is a depression assessment scale and contains 17 items pertaining to symptoms of depression experienced over the past week
The State and Trait Anxiety questionnaire | 4 weeks
  The State and Trait Anxiety questionnaire is has 20 items for assessing trait anxiety and 20 for state anxiety
The Korean Inventory of Depressive Symptomatology | 4 weeks
  The Korean Inventory of Depressive Symptomatology is a self-report questionnaire that comprises symptoms of depression including melancholic, atypical and anxious symptoms
The Perceived Stress Scale | 4 weeks
  The Perceived Stress Scale is is a measure of the degree to which situations in one's life are appraised as stressful
The Albany Panic and Phobia Questionnaire | 4 weeks
  The Albany Panic and Phobia Questionnaire is a 27-item 9-point Likert scale that was designed to measure the distinct dimension of fear in various situations, and has three subscales: social phobia, agoraphobia, and interoceptive fear
The Hospital Anxiety and Depression Scale | 4 weeks
  The Hospital Anxiety and Depression Scale is a 14-item scale that has anxiety and depression subscales;
The Body Sensations Questionnaire | 4 weeks
  The Body Sensations Questionnaire is a 17-item 5-point Likert scale that evaluates how afraid and anxious a patient is when he/she feels the physical sensation of each item in an unstable state
The Anxiety Sensitivity Index | 4 weeks
  The Anxiety Sensitivity Index is a 16-item measure tapping the fear of anxiety sensations, which is known to be a risk factor for the development of panic.

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Shin B, Oh J, Kim BH, Kim HE, Kim H, Kim S, Kim JJ. Effectiveness of Self-Guided Virtual Reality-Based Cognitive Behavioral Therapy for Panic Disorder: Randomized Controlled Trial. JMIR Ment Health. 2021 Nov 22;8(11):e30590. doi: 10.2196/30590. PMID 34813486